CLINICAL TRIAL: NCT05236543
Title: An Open-label, Fixed Sequence Study in Healthy Subjects to Assess the Pharmacokinetics of AZD4831 When Administered Alone and in Combination With Itraconazole
Brief Title: A Study to Assess the Pharmacokinetics of AZD4831 When Administered Alone and in Combination With Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6580C00013; 2021-005727-21 (EudraCT Number)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: Fixed Sequence Study; Cardiovascular Disease; Drug-drug interaction; Pharmacokinetics; Myeloperoxidase inhibitor
MeSH Terms: conditions — Cardiovascular Diseases | interventions — AZD4831; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive AZD4831 on Day 1; Itraconazole only on Days 8 through 10 , and AZD4831 and Itraconazole on Day 11 oral dosing of Itraconazole only on Days 12 through 17.
  Interventions: Drug: AZD4831; Drug: Itraconazole

INTERVENTIONS:
Drug: AZD4831 — Subjects will receive single oral dose only on Day 1 and Day 11.
Drug: Itraconazole — Subjects will receive Itraconazole orally on Days 8 followed by dosing from Day 9 to Day 17.

SUMMARY:
A study to demonstrate pharmacokinetics of AZD4831 when administered alone and in combination with Itraconazole.

DETAILED DESCRIPTION:
This will be a an open-label, 3-period fixed sequence study to be conducted at a single study centre.

The treatment starts with AZD4831 (Treatment Period 1), followed by Itraconazole administration for 3 days (Treatment Period 2) and finally a combination of AZD4831+Itraconazole administration (Treatment Period 3).

The study will comprise of:

* A Screening Period of approximately 28 days.
* Three Treatment Periods:

  * Treatment Period 1 (Day -1 through pre-dose Day 8): Single oral dose of AZD4831 only on Day 1,
  * Treatment Period 2 (Day 8 through pre-dose Day 11): Oral dose of Itraconazole only on Days 8 through 10,
  * Treatment Period 3 (Day 11 through Day 18, after the last PK sample is collected): AZD4831 and Itraconazole on Day 11 and oral dosing of Itraconazole only on Days 12 through 17.
* A final Follow-up Visit after the last PK sample (Day 25 to Day 32).

Each subject will be involved in the study for approximately 9 weeks (including the 28 day Screening Period).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female (non-childbearing potential) subjects aged 18 to 55 years (inclusive) at the time of signing informed consent, with suitable veins for cannulation or repeated venepuncture.
* Males must be willing to use appropriate contraception methods.
* Females must not be lactating and must be of non-childbearing potential.
* Have a .BMI between 18.5 and 30.0 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive) at Screening.

Exclusion Criteria:

* History of any clinically significant disease or disorder, including hyperthyroidism, uncontrolled hypothyroidism or any clinically significant thyroid disease.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational medicinal product (IMP).
* A positive COVID-19 test at the Screening Visit or admission to the Clinical Unit.
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis, vital signs, and 12-lead ECG.
* Any positive result at the Screening Visit for serum Hepatitis B surface antigen (HBsAg), HCV, and Human immunodeficiency virus (HIV) antibody.
* Known or suspected Gilbert's syndrome.
* Known or suspected history of drug abuse in the last 2 years, as judged by the Investigator.
* Has received another new chemical or biological entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study or final follow up visit within 1 month of first administration of IMP in this study.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to the Screening Visit.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4831 or itraconazole.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes).
* Excessive intake of caffeine-containing drinks or foods.
* Known or suspected history of alcohol or excessive intake of alcohol.
* Positive screen for drugs of abuse or cotinine at screening.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non prescribed medication including COVID-19 vaccines, antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life.
* Subjects who have previously received AZD4831.
* Subjects who are lactose intolerant or have other specific dietary restrictions that cannot be accommodated by the Clinical Unit.
* Subjects who, in the opinion of the Investigator, have any clinically significant skin condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Area under plasma concentration time curve from zero to infinity (AUCinf) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t½λz) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase (Vz/F) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Terminal elimination rate constant (λz) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRTinf) for AZD4831 | Period 1: Study days 1 to 6, 8; Period 3: Study days 11 to 16, 18
  To assess the effect of Itraconazole on AZD4831 only.

SECONDARY OUTCOMES:
Number of subjects with adverse events (AE) | From Screening (Day -28 to Day -2) to Follow-up visit (Between Day 25 and Day 32)
  To assess safety and tolerability of AZD4831 alone and in combination with Itraconazole.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home